CLINICAL TRIAL: NCT03870802
Title: Evaluation of Stem and Immune Cells in the Early Stage Breast Cancer Without Genetic Risk
Brief Title: MACSSI (MAstectomie Cellules Souches Surveillance Immunitaire)
Acronym: MACSSI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: MACSSI (ET18-150)
Record Dates: First submitted 2018-09-25; First posted 2019-03-12 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Stem cells; Immune cells
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breast tissue samples obtained during the prophylactic mastectomy
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Characterization of breast stem & immune system cells infiltrated in the mammary gland — Isolation, quantification and characterization of breast stem and immune cells of samples obtained during the prophylactic mastectomy in women presenting different tumor progression risks.

SUMMARY:
Monocentric, observational and prospective study in adult women having an early-stage breast cancer without genetic risk.

The main objective is to characterize quantitatively and qualitatively, after solitary confinement, the resident breast stem cells and the immune system cells infiltrated in the mammary gland in women:

* With a moderate risk of breast cancer progression (women with an early "Luminal A" tumor) = Group A.
* With a high risk of breast cancer progression (women with an early "Luminal B" or basal tumor) = Group B.

DETAILED DESCRIPTION:
Breast cancer is one of the most frequent and the second cause of mortality for women in the world. Breast is a complex organ which has several changes (puberty, pregnancy and menopause). These modifications are controlled by numerous signals as those transmitted by the oestrogens. They are possible through the presence of stem cells in the mammary gland which are able to reply to these signals and can be the target of alterations leading to cancer cells occurence. Breast tumors are composed of complex entities of different kinds of cancer and normal cells which constitute the tumor micro-environment including the immune system cells. This micro-environment transmits a lot of signals to cancer cells and particularly stem cells which can contribute to their survival, the tumor progression and interfere with the treatments efficacy.

The detection of the major deregulation of BMP2 synthesis by mammary micro-environment cells may be a reliable and early biomarker of carcinogens exposure and an indicator of a high risk of developing a luminal type breast cancer.

The immune micro-environment, which has an impact on solid cancer patients' survival, should be taken into consideration for new therapeutic strategies.

Some infiltrating tumour immune cells, as macrophages (TAM) or regulating T and B cells, have shown their key role in tumour escape and metastases apparition. It is relevant to associate the evaluation of immune infiltrate to the breast stem cells in early stage tumours since the literature suggests a functional interaction of these two cellular compartments, particularly in the glioblastoma and the prostate cancer. It seems that mammary stem cells are a major element in the comprehension of breast carcinogenesis but also in the possibilities of repairing the mammary tissue controlling the mammary carcinogenesis.

It is fundamental to clarify the role of stem cells and immunity. Our hypothesis is that breast stem cells are altered in women having a high risk of cancer progression. They would be responsible for a reduced activity of cellular repair and/or contribute to tumour development.

MACSSI project consists in isolating, quantifying and characterizing the breast stem cells and the isolated immune cells of samples obtained for the prophylactic mastectomy in women presenting different tumour progression risks.

The results will be compared to normal samples already collected in women who had a breast reduction.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient requiring a breast surgery (total mastectomy) of an early stage tumour classified as :

  * Luminal A (Arm A) : Patients with a moderate risk of breast cancer progression or,
  * Luminal B or Basal (Arm B) : Patients with a high risk of breast cancer progression
* Systemic treatment not initiated
* Breast cup size ≥ C
* Informed and signed consent.

Exclusion Criteria:

* Neo-adjuvant chemotherapy or hormonotherapy
* History of breast irradiation
* Pregnant or breastfeeding woman
* Patient under tutorship or curatorship
* Patient who underwent a lumpectomy with a level-2 oncoplastic surgery (ex: breast reduction with an inverted-T remodeling)
* Any other prior anti-tumor treatment
* Other medical pathology which may interfere with the biologic evaluation, especially chronic auto-immune diseases.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult women having an early-stage breast cancer without genetic risk
Study Population: Adult women having an early-stage breast cancer without genetic risk requiring a breast surgery
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-02-22 (Actual); Primary Completion 2024-02-22 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
To characterise quantitatively and qualitatively, after solitary confinement, the resident breast stem cells and the immune system cells infiltrated in the mammary gland according to the risk of breast cancer progression (group A and B) | Within one month after inclusion (date of surgery)
  Rate of stem and immune cells and phenotype analysis

SECONDARY OUTCOMES:
Functional characterization, after solitary confinement, of stem cells and immune system cells from groups A and B | Within one month after inclusion (date of surgery)
  Functional test: mammosphere
Functional characterization, after solitary confinement, of stem cells and immune system cells from groups A and B | Within one month after inclusion (date of surgery)
  Functional test: TDLU
Functional characterization, after solitary confinement, of stem cells and immune system cells from groups A and B | Within one month after inclusion (date of surgery)
  Functional test: E-CFC - FACS
Determination of the stem cells role in the cellular regulation and repair activity | Within one month after inclusion (date of surgery)
  Functional tests
Determination of the efficacy of the immune systems cells found in the samples in the early stage of breast tumorigenesis | Within one month after inclusion (date of surgery)
  FACS
Evaluation of the role of breast stem and immune cells in the early stage development of a breast cancer: risk or protective factor ? | Within one month after inclusion (date of surgery)
  Functional tests: mammosphere, TDLU, E-CFC - FACS

CONTACTS AND LOCATIONS:
Overall Officials: DELAY Emmanuel, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France